CLINICAL TRIAL: NCT05733988
Title: Edge-To-Edge Technique Used as a Bailout in Case of Sub-Optimal Mitral Repair: Very Long-Term Results
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: ETEB-SOR-VLT
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bailout edge to edge — Edge to edge repair is the suture of the mitral valve leaflets in the regurgitant spot. It can be used as a bailout procedure when the first attempt of mitral valve repair with other surgical techniques is not satisfactory at intraoperative echo control. In this case, a second run of cardiopulmonary bypass is carried out, the heart is reopened and an edge-to-edge is performed.

SUMMARY:
The absence of residual mitral regurgitation (MR) after mitral valve repair is of paramount importance for the long term durability of the valve repair. Thus, ideally, after weaning from cardio-pulmonary by-pass (CPB) the trans-esophageal echocardiogram (TEE) should show no (or only trivial) residual MR, good coaptation length and no iatrogenic mitral valve stenosis. However, mild or more residual MR can be present in up to 4% of the patients after the initial mitral valve repair and a second CPB run may be necessary to improve the repair results. Mechanism of residual MR can be dynamic, related to systolic anterior motion (SAM) or to severe left ventricular dysfunction, and anatomical, related to residual prolapse, cleft, and suture or ring dehiscence. In several cases medical therapy can be effective in the management of the intra-operatively detected SAM, and residual cleft or suture dehiscence can be easily corrected during a second CPB run. However, in other cases SAM is not responsive to medical therapy or the residual MR jet would require complex and time-consuming techniques to be addressed, or even worse scenario, a mitral valve replacement could be necessary. In such cases the edge-to-edge (EE) technique can be used as a bail-out procedure. The anatomical characteristics of the mitral valve after an initial sub-optimal repair are certainly not ideal for the edge-to-edge technique, due to a possible significant reduction in the valve area, especially in case of posterior leaflet resection or small ring implanted. Nevertheless, in the short term the edge-to-edge technique used to rescue patients with sub-optimal initial repair resulted effective. However, the very long-term results of the edge-to-edge technique used as bail-out are not known. Thus, the aim of this study is to evaluate the clinical and echocardiographic results of the edge-to-edge technique used to rescue patients with initial sub-optimal mitral repair.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Patients underwent mitral valve repair, with more than mild residual MR at the intraoperative TEE after leaving the CPB;
* Patients in whom EtE alone has been added to the repair already performed, as a technique to reduce residual MR after first attempt of mitral valve repair;
* Patients operated both in median sternotomy or in minithoracotomy;
* Patients operated on at the Cardiac Surgery departmet of San Raffaele Hospital since January 1999 to December 2015.

Exclusion Criteria:

* Patients in whom other techniques have been used as a bailout procedure, concurrently or instead of EtE;
* Patients where the initial repair has been modified or undone;
* Patients whose mitral valve has been replaced.

Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a mitral valve repair surgery and in whom, at the intraoperative echo control, results where not satisfying, so an edge-to-edge repair was also performed as a bailout procedure
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 22 years
Reintervention for MR recurrency | Up to 22 years
MR recurrency | Up to 22 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No